CLINICAL TRIAL: NCT05261633
Title: Diffusion Magnetic Resonance Imaging (MRI) of the Abdomen
Brief Title: Diffusion MRI of the Abdomen
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2021-1289; Protocol Version 10/17/2025 (Other: UW Madison); A539300 (Other: UW Madison); 1R01EB030497-01 (NIH)
Record Dates: First submitted 2022-02-03; First posted 2022-03-02 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Abdominal Imaging
MeSH Terms: interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Healthy Volunteers
  Interventions: Device: Diffusion Weighted Magnetic Resonance Imaging
- Known Liver Metastases
  Interventions: Device: Diffusion Weighted Magnetic Resonance Imaging

INTERVENTIONS:
Device: Diffusion Weighted Magnetic Resonance Imaging — Diffusion-weighted (DW)-MRI has a unique ability to probe tissue microstructure without the need for ionizing radiation or intravenous contrast agents. DW-MRI of the abdomen is utilized in detection, staging, and treatment surveillance of malignancies, and has shown great promise in various other applications, including for the assessment of fibrosis in the liver, pancreas, kidneys, and other organs.
  Other Names: DW-MRI

SUMMARY:
The purpose of this research is to see if a new magnetic resonance imaging (MRI) method will be able to improve the images taken of the abdomen. This new method includes some changes to help avoid movements that may disrupt the images like breathing, heartbeats and other involuntary motion that occurs in the abdomen. This study will these methods in healthy volunteers and validate them in patients with known liver metastases in a single contrast-enhanced MRI visit.

DETAILED DESCRIPTION:
This study will develop and validate novel DW-MRI methods with unprecedented robustness to motion, favorable image quality, and quantitative precision for abdominal imaging. Upon successful completion, these methods will have broad applications, including the assessment of cancer, fibrosis and other disease processes in various abdominal organs such as the liver, pancreas, kidneys, bowel and beyond.

The primary objective is to demonstrate precise quantitative diffusion parameter mapping that is achieved by the novel, motion-robust, low-distortion DW-MRI methods in a representative and clinically relevant application, for the assessment of liver metastatic disease. Specifically, the investigators will:

1. Compare the repeatability of DW-MRI methods by calculating the squared difference between each pair of repeated ADC measurements in lesions and healthy tissue, and will model this value including the DW-MRI method as a covariate using Generalized Estimating Equations (GEE).

Secondary objectives include optimization of the methods in healthy volunteers, assessment of image quality and distortions, as well gathering preliminary data for assessment of sensitivity and specificity for detection of lesions:

1. Optimization in healthy volunteers

   1. (Aim 1) Optimized bh, M1 and M2 parameters by minimization of the mean squared error and bias of ADC quantification across the liver
   2. (Aim 2) Optimized motion-corrected averaging via image quality assessment by three radiologists using a Likert scale.
2. SNR (signal-to-noise ratio) will be evaluated for each DW-MRI dataset, using an expectation-maximization method, accounting for parallel imaging, spatially varying noise, and magnitude operation.
3. To assess image distortions in DW-MRI, the cross-correlation coefficient (CCC) will be used to assess alignment between each of the DW-MRI datasets and the reference T2-weighted acquisition.
4. Each DW-MRI reconstruction will be evaluated by three radiologists using a Likert scale between 0 (worst/non-diagnostic) and 4 (best) for several criteria: motion artifacts, spatial resolution, distortions, apparent SNR, and overall image quality. The post-contrast images will serve as a guide to assess for artifacts by demonstrating the liver and the lesions.
5. Per-lesion sensitivity, specificity, and accuracy will be assessed for each DW-MRI method. McNemar's test will be used to compare the sensitivity and specificity between methods.
6. Intra-reader variability will be assessed by each reader will repeating ADC measurements after two months.
7. Inter-reader variability will be assessed in ADC measurements by comparing matching lesions, based on the recorded lesion location across readers.

Specific Aims Aim 1: Optimize a reliable, motion-robust DW-MRI of the abdomen in healthy volunteers.

Aim 2: Optimize, in healthy volunteers, a high-resolution, low-distortion, motion-robust DW-MRI of the abdomen through the synergistic combination of motion-robust DW-MRI with state-of-the-art low-distortion techniques.

Aim 3: Demonstrate excellent image quality and precise quantitative diffusion parameter mapping using the novel DW-MRI methods in a representative and clinically relevant application for the assessment of liver metastases, by evaluating in patients:

3a. Quantitative and subjective image quality metrics. 3b. Precision (test-retest repeatability) of ADC measurements in the liver (including healthy parenchyma and lesions) by novel vs. standard DW-MRI methods.

ELIGIBILITY:
Inclusion Criteria for Healthy Volunteers:

* 18 years of age or older

Exclusion Criteria for Healthy Volunteers:

* Patients with contraindication to MRI (e.g. pacemaker, contraindicated metallic implants, claustrophobia, etc)
* Pregnant or trying to become pregnant (as determined by self-report during MRI safety screening)

Inclusion Criteria for Patients:

* 18 years of age or older
* Patients with at least one of the following:

  * Radiologically visible solid tumor liver metastasis, with at least one metastatic liver lesion must be a minimum of 8 mm in longest diameter
  * Patients presenting for liver lesion biopsy

Exclusion Criteria for Patients:

* Patients with contraindication to MRI (e.g. pacemaker, contraindicated metallic implants, claustrophobia, etc)
* Patients with known contraindication to GBCA such as severe kidney disease or previously documented GFR < 30 ml/min/1.73 m2
* Patients requiring intravenous (IV) conscious sedation for imaging are not eligible; patients requiring mild, oral anxiolytics for the MRI will be allowed to participate as long as the following criteria are met:

  * The subject has their own prescription for the medication.
  * The informed consent process is conducted prior to the self-administration of this medication
  * They come to the research visit with a driver
* Pregnant or trying to become pregnant (as determined by self-report during MRI safety screening)
* Stent in bile ducts
* Partial hepatectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and people with known liver metastases that are 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Squared difference between each pair of repeated ADC measurements | up to 1.5 hours
  Compare the repeatability of DW-MRI methods by calculating the squared difference between each pair of repeated apparent diffusion coefficient (ADC) measurements in lesions and healthy tissue, and will model this value including the DW-MRI method as a covariate using Generalized Estimating Equations (GEE).

SECONDARY OUTCOMES:
Mean Squared Error of ADC in images from Healthy Volunteers | up to 1.5 hours
  Optimized bh, M1 and M2 parameters in healthy volunteers by minimization of the mean squared error and bias of ADC quantification across the liver.
Image Quality Score in images from Healthy Volunteers | up to 1.5 hours
  Optimized motion-corrected averaging in healthy volunteers via image quality assessment by three radiologists using a Likert scale, ranging between 0 (worst/non-diagnostic) and 4 (best).
Signal-to-Noise Ratio (SNR) | up to 1.5 hours
  SNR will be evaluated for each DW-MRI dataset, using an expectation-maximization method, accounting for parallel imaging, spatially varying noise, and magnitude operation
Cross-correlation coefficient (CCC) of images | up to 1.5 hours
  To assess image distortions in DW-MRI, the cross-correlation coefficient (CCC) will be used to assess alignment between each of the DW-MRI datasets and the reference T2-weighted acquisition.
Overall Image Quality Score | up to 1.5 hours
  Each DW-MRI reconstruction will be evaluated by three radiologists using a Likert scale between 0 (worst/non-diagnostic) and 4 (best) for several criteria: motion artifacts, spatial resolution, distortions, apparent SNR, and overall image quality. The post-contrast images will serve as a guide to assess for artifacts by demonstrating the liver and the lesions.
Sensitivity: Number of True Positive Assessments divided by Number of All Positive Assessments | up to 1.5 hours
  Per-lesion sensitivity will be assessed for each DW-MRI method. McNemar's test will be used to compare the sensitivity and specificity between methods.
Specificity: Number of True Negative Assessments divided by Number of All Negative Assessments | up to 1.5 hours
  Per-lesion specificity will be assessed for each DW-MRI method. McNemar's test will be used to compare the sensitivity and specificity between methods.
Accuracy: Number of Correct Assessments divided by Number of All Assessments | up to 1.5 hours
  Per-lesion accuracy will be assessed for each DW-MRI method. McNemar's test will be used to compare the sensitivity and specificity between methods.
Repeat ADC Measurements to Assess Intra-Reader Variability | up to 1.5 hours
  Intra-reader variability will be assessed by each reader with repeating ADC measurements after two months
ACD Measures For Each Reader to assess Inter-Reader Variability | up to 1.5 hours
  Inter-reader variability will be assessed in ADC measurements by comparing matching lesions, based on the recorded lesion location across readers.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Hernando, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No